CLINICAL TRIAL: NCT01934218
Title: A Multi-Center, Randomized, Double-Blind, Phosphate Buffered Saline-Controlled Study to Evaluate Effectiveness and Safety of a Single Intra-Articular Injection of Gel-One® for the Treatment of Osteoarthritis of the Knee With Open-Label Safety Extension
Brief Title: Gel-One Treatment in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seikagaku Corporation (Industry)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gel/1133
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Osteoarthritis Knee
Keywords: Knee; Osteoarthritis; Intra-articular injection
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gel-One (Active Comparator): 3 mL, a single intra-articular injection of Gel-One
  Interventions: Device: Gel-One
- Phosphate Buffered Saline (PBS) (Placebo Comparator): 3 mL, a single intra-articular injection of PBS
  Interventions: Device: PBS

INTERVENTIONS:
Device: Gel-One
  Arms: Gel-One
Device: PBS
  Arms: Phosphate Buffered Saline (PBS)

SUMMARY:
The purpose of this study is to determine whether Gel-One demonstrates a superior effectiveness in osteoarthritis (OA) knee pain compared with phosphate buffered saline (PBS) injections.

ELIGIBILITY:
Inclusion Criteria:

* Have a knee pain
* Grade 1 to 3 on the Kellgren-Lawrence grading scale

Exclusion Criteria:

* BMI greater than 35 kg/m2
* Received an intra-articular hyaluronic acid injection for the treatment of OA of the knee within 6 months prior to screening
* Had a joint replacement of the target knee

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 814 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - Birmingham, Alabama
  - Sheffield, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Cerritos, California
  - Costa Mesa, California
  - Garden Grove, California
  - North Hollywood, California
  - San Diego, California
  - Boulder, Colorado
  - Englewood, Colorado
  - Cos Cob, Connecticut
  - Trumbull, Connecticut
  - Oviedo, Florida
  - Pinellas Park, Florida
  - Plantation, Florida
  - Sarasota, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - Marietta, Georgia
  - Morton Grove, Illinois
  - Newton, Kansas
  - Wichita, Kansas
  - Lake Charles, Louisiana
  - Wheaton, Maryland
  - St Louis, Missouri
  - Trenton, New Jersey
  - Hartsdale, New York
  - New York, New York
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Altoona, Pennsylvania
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - State College, Pennsylvania
  - Austin, Texas
  - Bedford, Texas
  - Charlottesville, Virginia

REFERENCES:
- [Derived] Takamura J, Seo T, Strand V. A Single Intra-Articular Injection of Gel-200 for Treatment of Symptomatic Osteoarthritis of the Knee Is More Effective than Phosphate Buffered Saline at 6 Months: A Subgroup Analysis of a Multicenter, Randomized Controlled Trial. Cartilage. 2019 Oct;10(4):417-422. doi: 10.1177/1947603518768015. Epub 2018 Apr 12. PMID 29644875

RESULTS

PARTICIPANT FLOW:
Groups:
- Gel-One: The participants received a single intra-articular injection of Gel-One.
- Placebo: The participants received a single intra-articular injection of Phosphate Buffered Saline (PBS).
Period: Double-blind Phase
Arm/Group | Gel-One | Placebo
Started | 404 | 410
Analyzed Participants (5 subjects removed from ITT analyses because of no post treatment data. (Pre-defined)) | 402 | 407
Completed | 356 | 356
Not Completed | 48 | 54
Not completed — Adverse Event | 8 | 8
Not completed — Lack of Efficacy | 6 | 7
Not completed — Lost to Follow-up | 7 | 14
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 4 | 0
Not completed — Withdrawal by Subject | 16 | 13
Not completed — Noncompliance with Study Protocol | 5 | 8
Not completed — Protocol Violation of Study Eligibility | 1 | 2
Period: Open-Label Phase
Arm/Group | Gel-One | Placebo
Started | 316 | 328
Completed | 290 | 304
Not Completed | 26 | 24
Not completed — Adverse Event | 2 | 4
Not completed — Lack of Efficacy | 1 | 4
Not completed — Lost to Follow-up | 4 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 13 | 11
Not completed — Noncompliance with Study Protocol | 4 | 2
Not completed — Failure to Exam Primary Evaluation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: The participants received a single intra-articular injection of PBS.
- Total: Total of all reporting groups
Arm/Group | Gel-One | Placebo | Total
Number analyzed (Participants) | 402 | 407 | 809
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (9.14) | 59.8 (9.32) | 59.6 (9.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221 | 234 | 455
  Male | 181 | 173 | 354
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 28 | 63
  Not Hispanic or Latino | 367 | 379 | 746
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 52 | 52 | 104
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 93 | 70 | 163
  White | 247 | 277 | 524
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 7 | 17
Body mass index [Mean (Standard Deviation); unit: kilograms / meter square] | 28.597 (4.1923) | 28.797 (3.9244) | 28.698 (4.0585)
Kellgren-Lawrence score [Number; unit: participants] — The Kellgren-Lawrence score is radiological classification of knee osteoarthritis. It progresses from grade 0 to grade IV and classified based on x-rays.
  participants
    1 | 113 | 111 | 224
    2 | 161 | 164 | 325
    3 | 128 | 132 | 260
osteoarthritis knee disease duration [Mean (Standard Deviation); unit: years] | 6.80 (7.835) | 6.90 (7.072) | 6.85 (7.456)
Etiology [Number; unit: participants]
  Idiopathic | 359 | 359 | 718
  Post-traumatic | 43 | 48 | 91
Study knee [Number; unit: participants]
  Right | 209 | 212 | 421
  Left | 193 | 195 | 388
50-foot walk test VAS pain score [Mean (Standard Deviation); unit: mm] — Observed Visual Analogue Scale (VAS) pain score of 100 mm; 0 mm meaning no pain; 100 mm meaning extreme target knee pain following 50-foot walk test.
  mm | 69.25 (7.640) | 69.36 (7.817) | 69.31 (7.725)
50-foot walk test contralateral VAS pain score [Mean (Standard Deviation); unit: mm] — Observed VAS pain score of 100 mm; 0 mm meaning no pain; 100 mm meaning extreme contralateral knee pain following 50-foot walk test.
  mm | 11.50 (7.536) | 11.95 (7.565) | 11.73 (7.549)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Visual Analogue Scores (VAS) Following 50-foot Walk Test Through Week 26
Description: Observed VAS of 100 mm; 0 mm meaning no pain; 100 mm meaning extreme pain following 50-foot walk test. Change in score from baseline through week 26 was estimated using a longitudinal model.
Time Frame: Baseline up to Week26
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Gel-One | Placebo
Number analyzed (Participants) | 402 | 407
mm | -31.7 [-33.7 to -29.6] | -31.7 [-33.7 to -29.6]
Statistical Analysis 1: Comparison: Gel-One vs Placebo; Test type: Superiority; p = 0.988, Basic longitudinal model; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-2.7 to 2.7]

2. Post Hoc Outcome: Change From Baseline in Visual Analogue Scores (VAS) Following 50-foot Walk Test at Week 26
Description: Observed VAS of 100 mm; 0 mm meaning no pain; 100 mm meaning extreme pain following 50-foot walk test. Change in score from baseline to week 26 was calculated as baseline minus week 26.
Time Frame: Baseline and Week 26
Population: The post-hoc analysis plan pre-specified that only the change at week 26 in the Gel-One arm is intended to be analyzed.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Gel-One
Number analyzed (Participants) | 402
mm | -29.5 [-32.1 to -26.9]
Statistical Analysis 1: Comparison: Gel-One; A post-hoc non-inferiority comparison of the Gel-One mean change from baseline in VAS pain score at week 26 (Following 50-foot walk test) against the same assessment collected from subjects treated with Euflexxa in a separate study (PMID:19539353) was also performed; Test type: Other — Euflexxa would be considered superior to Gel-One if the difference in mean change from baseline in VAS pain score at week 26 was 5 mm or greater (on the 100mm VAS pain scale). If the difference in mean change values were within 5 mm, Gel-One would not be considered inferior to Euflexxa; Change from baseline (95% CI) for Euflexxa was -25.7 (-29.0, -22.4) and the difference between Euflexxa and Gel-One (95% CI) was -3.8 (-inf, -0.3)

ADVERSE EVENTS:
Time Frame: 25 months
Groups:
- Placebo: 3 mL, a single intra-articular injection of PBS.
Arm/Group | Gel-One | Placebo
All-Cause Mortality (participants affected / at risk) | 0/404 | 0/410
Serious Adverse Events (participants affected / at risk) | 7/404 | 6/410
Other Adverse Events (participants affected / at risk) | 107/404 | 113/410
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gel-One (N=404) | Placebo (N=410)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gel-One (N=404) | Placebo (N=410)
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 | 42
Joint swelling (Musculoskeletal and connective tissue disorders) | 33 | 42
Joint effusion (Musculoskeletal and connective tissue disorders) | 30 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other